CLINICAL TRIAL: NCT03500666
Title: A Comparative Study of Robot Assisted BABA Approach and Chest Breast Approach for Lateral Neck Dissection
Brief Title: Comparative Study of Robot BABA Approach and Chest Breast Approach for Lateral Neck Dissection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Bo Wang,MD, clinical professor, Fujian Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BND and RND
Record Dates: First submitted 2018-04-02; First posted 2018-04-18 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Thyroid Carcinoma; Robot Surgery; Endoscopic Surgery
Keywords: Thyroid carcinoma; Robot surgery; Endoscopic surgery
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Robotic Surgical Procedures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robot lateral neck lymph node dissection (Experimental): Robot neck lateral lymph node dissection was performed in patients with thyroid cancer and lateral cervical lymph node metastasis.
  Interventions: Device: Robot
- Total endoscopic lateral cervical lymph node dissection (Experimental): Patients with thyroid cancer and lateral cervical lymph node metastases underwent total endoscopic neck dissection.
  Interventions: Device: Total endoscopic

INTERVENTIONS:
Device: Robot — Robot lateral neck lymph node dissection
  Other Names: Robot lateral neck lymph node dissection
  Arms: Robot lateral neck lymph node dissection
Device: Total endoscopic — Total endoscopic lateral cervical lymph node dissection
  Other Names: Total endoscopic lateral cervical lymph node dissection
  Arms: Total endoscopic lateral cervical lymph node dissection

SUMMARY:
Objective to compare the advantages and disadvantages of robotic and conventional endoscopic thyroidectomy for thyroid cancer.

DETAILED DESCRIPTION:
To compare the difference of operative time and complication between two operative methods in robot neck surgery and routine endoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

1. papillary thyroid carcinoma with clinically suspected or confirmed lateral lymph node metastasis;
2. patient's concerns of neck scars and cosmetic requirement.

The exclusion criteria were as follows:

1) tumor size >4cm; 2) previous neck surgical history； 3）residual or recurrent tumors; 4) suspicious primary tumor or metastatic lymph node invasion of major vascular structures or recurrent laryngeal nerve.

5）metastatic lymph nodes occurred below the sternoclavicular joint.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Lateral cervical lymph node cleaning time | During surgery
  Lateral cervical lymph node clean time from that beginning of cut the SCM leading edge to the end of the specimen
Accessory nerve injury | During surgery
  Accessory nerve injury
Intraoperative internal jugular vein bleeding. | 6 months after surgery
  Internal carotid vein hemorrhage affect that surgical procedure

SECONDARY OUTCOMES:
The time of the thyroid gland removal | During surgery
  The time of the thyroid gland removal , including the opening of the white line to the thyroid, and the end of the specimen
Number of participants with HypoParathyroidism | 6 months after surgery
  The parathyroid function was examined six months after surgery.
Recurrent laryngeal nerve injury. | 6 months after surgery
  The recurrent laryngeal nerve function due to nerve injury or thermal damage can not be recovered for 6 months.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Wen-xin ZHAO, Fuzhou, Fujian

IPD SHARING:
Plan to Share IPD: No